CLINICAL TRIAL: NCT04567277
Title: Early Ventriculo-peritoneal Shunt in Subarachnoid Patients With External Ventricular Drainage
Acronym: EarlyVPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mashhad University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Humain Baharvahdat, Neurosurgical Department, Mashhad University of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T5097
Record Dates: First submitted 2020-09-23; First posted 2020-09-28 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Subarachnoid Hemorrhage; Ventriculo-Peritoneal Shunt Infection; Hydrocephalus
Keywords: High grade subarachnoid hemorrhage; External ventricular drainage; Ventricular-peritoneal shunt
MeSH Terms: conditions — Subarachnoid Hemorrhage; Hydrocephalus

STUDY DESIGN:
Intervention Model Description: The study has a single group including patients with high grade subarachnoid hemorrhage (WFNS 3-4) for whom EVD was inserted. EVD was tried converted into VPS within 7-10 days of insertion.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Early VPS (Experimental)
  Interventions: Procedure: External ventricular drainage (EVD) conversion into ventriculo-peritoneal shunt (VPS)

INTERVENTIONS:
Procedure: External ventricular drainage (EVD) conversion into ventriculo-peritoneal shunt (VPS) — EVD in high grade SAH patients were converted into VPS with 7-10 days of EVD insertion

SUMMARY:
Acute hydrocephalus is a common complication following subarachnoid hemorrhage (SAH). Early and emergency insertion of external ventricular drain (EVD) is standard treatment of acute post-SAH hydrocephalus. According to the high risk of infection associated with EVD, the study evaluates the outcome of early EVD conversion to ventriculoperitoneal shunt (VPS) in poor-grade SAH patients.

DETAILED DESCRIPTION:
This study was performed on patients diagnosed with high grade SAH (WFNS 4-5) who undergo EVD within 24 hours of their admission. The conversion of EVD to VPS is performed within 7-10 days of EVD insertion, defined as early VPS group. The ventricular catheter is inserted in lateral ventricle using the same burr hole of EVD or the contralateral Kocher's point. All ruptured aneurysms could be closed by endovascular techniques or surgery.

The goal is to discontinuing EVD or its conversion to VPS within 7 to 10 days of insertion. At day 5-7 of EVD insertion, the EVD level is elevated from 15 cmH2O to 25 centimeter of water (cmH2O) gradually. The patients is evaluated during the 48 hours for cerebrospinal fluid (CSF) volume discharge, neurological consciousness, and hydrocephalus within brain CT scan acquired at the end of 48 hours of observation. If the daily CSF fluid discharge will be greater than 100 ml, brain CT scan shows evidence of HCP, there is any CSF leak from around the catheter, or the patient experiences GCS drop for 2 points or more, EVD is converted to VPS.

EVD conversion to VPS is postponed if there is any evidence of CSF infection within the last CSF analysis obtained 48 hours before VPS placement, patient experiences fever (>38.5° C) without any other source, or there is any evidence of severe vasospasm in transcranial Doppler (TCD) imaging or brain CT angiography. Otherwise, The EVD is discontinued.

For all patients, a brain CT scan is taken to evaluate the location of shunt 24 hours after VPS placement. Forty-eight hours after VPS placement, lumbar puncture (LP) is performed to collect CSF for ruling out the possibility of shunt infection or ventriculitis. Shunt malfunction (approved by imaging or signs of HCP) is reported if it occurred within 3 months of VPS placement.

When VPS malfunction is diagnosed it is revised. CSF infection is considered if there is a positive culture or ratio of CSF white blood cell count (WBC)/ red blood cell count (RBC) to blood WBC/RBC was more than 3. All patients is evaluated for clinical condition using modified Rankin scale (mRs) at discharge and 6 months later.

ELIGIBILITY:
Inclusion Criteria:

* patients with SAH and World Federation of Neurosurgeon (WFNS) Grade 4 or 5 and
* patient who underwent ventriculostomy (EVD insertion) within 24 hours of SAH onset.

Exclusion Criteria:

* patients with Glasgow Coma Scale of (GCS) 3 and fixed non-reactive pupils,
* patients in whom EVD was inserted in the other hospital,
* patients were successfully weaned from EVD with 7-10 days of EVD insertion
* patients who died during hospitalization.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2021-02 (Actual); Study Completion 2021-03 (Actual)

PRIMARY OUTCOMES:
rate of ventriculo-peritoneal malfunction | 3 months
  VPS is defined malfunction when signs of hydrocephalus are seen in imaging (CTS or MRI)/clinical findings
rate of ventricle-peritoneal infection | 3 months

SECONDARY OUTCOMES:
RBC / protein level in CSF association with VPS malfunction | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Ghaem Hospital, Mashhad University of Medical Sciences, Mashhad, Iran

IPD SHARING:
Plan to Share IPD: Undecided